CLINICAL TRIAL: NCT04350346
Title: A Prospective, Randomized Controlled Trial of the Comparative Analysis Between Motilitone and Gasmotin for the Symptom Relief in Gallstone Patients With Functional Dyspepsia
Brief Title: The Comparative Analysis Between Motilitone and Gasmotin for the Symptom Relief in Gallstone Patients With Functional Dyspepsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 4-2019-0728
Record Dates: First submitted 2020-04-08; First posted 2020-04-17 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Gallstone
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The patient group who taken Motilitone (Active Comparator)
  Interventions: Drug: Motilitone
- The patient group who taken Gasmotin (Active Comparator)
  Interventions: Drug: Gasmotin

INTERVENTIONS:
Drug: Motilitone — 1. Ingredients and content: corydalis tuber, pharbitis seed 50% EtOH extracts 30mg
  2. Dosage method: Usually, adults take 1 tablet 3 times a day orally before meals.
  3. Pharmacological action:
     * It stimulates 5-HT4 receptor as a gastrointestinal motility accelerator to increase acetylcholine secretion and contract smooth muscle.
       * Stimulates stomach smooth muscle contraction by suppressing the effect of dopamine on acetylcholine secretion by inhibiting D2 receptor ③ It shows a pharmacological action that stimulates gastrointestinal movement by acting in combination with 5-HT1A / B receptor.
  Arms: The patient group who taken Motilitone
Drug: Gasmotin — 1. Ingredient and content: mosapride citrate dihydrate 5.29mg (5mg as active ingredient)
  2. Dosage method: Usually, an adult is orally administered 1 tablet 3 times a day before meals.
  3. Pharmacological action: mosapride is a selective serotonin-4 (5-HT4) receptor agonist with gastrointestinal stimulating activity, contracting smooth muscle
  Arms: The patient group who taken Gasmotin

SUMMARY:
* (Cause of cholelithiasis) Recently, the average age has increased, and the occurrence of gallstones has increased as the dietary life has been westernized due to the improvement of socio-economic level. When cholesterol increases, the occurrence of gallstones increases. Factors include high-calorie high-fat diet, increasing age, women, pregnant women, obesity, and oral contraceptives. There are cases. As another cause, gallstones occur well even when bile stasis occurs due to a decrease in motility of the gallbladder. These are conditions that lower mobility. And cholelithiasis has a genetic tendency in about 30%. In addition, since the eating habits of the family are similar, the genetic factors and the eating habits overlap, which often leads to the occurrence of cholelithiasis in the family.
* (symptoms of cholelithiasis) In most cases, complaints of non-specific digestive system symptoms, such as abdominal bloating, nausea, and especially indigestion after fatty diet, are often observed. According to domestic reports, the nonspecific symptoms complained by patients with cholelithiasis were indigestion, flatulence, frequent belching, nausea, loss of appetite, diarrhea, and vomiting. In general, many healthy people without gallstones complain of non-specific digestive system symptoms in 50% of cases, and there is a possibility that functional gastrointestinal diseases such as dyspepsia, peptic ulcer, and gastritis may be accompanied by these digestive system symptoms. It is difficult to know whether it is unrelated to gallstones. Symptoms caused by typical cholelithiasis usually have a characteristic that they often improve on their own after a few hours, and the start and end of the symptoms are relatively clear and repeatedly occur. In addition, various symptoms are displayed depending on the presence or absence of inflammation and progression.
* (Principle of treatment of cholelithiasis)

  1. Medical treatment: Medical treatment of gallstones is a method of dissolving using drugs to treat cholesterol gallstones in gallbladder stones. In 1973, Nakano et al. [1] published the first example of dissolving cholesterol gallstones using ursodeoxycholic acid (UDCA). Currently, UDCA is the only drug administered to patients with asymptomatic or mild symptoms of cholelithiasis in actual clinical practice, and there is no specific prescription drug.
  2. Surgical treatment: In the case of indications of cholecystectomy, acute cholecystitis, severe symptoms, chronic cholecystitis with severe thickening of the gallbladder wall, repeated and severe symptoms, porcelain gallbladder, Patients with gallstones of 3 cm or more in size, patients with anomalous pancreato-biliary duct unions, or gallbladder polyps.
* (Study on increasing gallbladder contractility) So far, there have been studies that some drugs increase or decrease gallbladder contractility. Catnach SM et al. [2] reported that erythromycin increased gallbladder contractility in patients with autonomic neuropathy due to diabetes. Sengupta S et al. [3] reported that indoramin (α-adrenergic antagonist), a prokinetic agent, increased gallbladder contractility in patients with cholelithiasis, resulting in a significant decrease in gallbladder volume.

Motilitone® developed in Korea is a gastrointestinal motility stimulator that stimulates 5-HT4 receptors to increase acetylcholine secretion and has a mechanism of contracting smooth muscles, improving symptoms in patients with functional dyspepsia in cholelithiasis It is expected to be able to give, and it is thought to have the effect of preventing the crystallization of bile acids due to an increase in the gallbladder contractility, thereby preventing the formation of gallstones and preventing newly generated gallstones.

To date, there are no special drugs for dyspepsia or pain improvement in patients with cholelithiasis. It is hypothesized that administration of motilitone® will increase the contractile capacity of the gallbladder, thereby improving digestion and preventing further formation of gallstones. As a control group, Gasmotin® was administered to improve functional dyspepsia, and the degree of symptom improvement was measured and compared by completing the Symptom Score Questionnaire for Indigestion between the two groups.

DETAILED DESCRIPTION:
At Severance Hospital, patients with cholelithiasis with symptoms of indigestion are divided into the Motilitone® and Gasmotin® groups. Provide sufficient oral and written explanation of the clinical trial and obtain consent from the patient who has revealed his willingness to participate. Randomization uses random numbers, and patient assignment by random numbers is managed by a third party who does not have direct contact with the patient or clinical history, and after obtaining consent, the group according to the random number is given and medication is given. It is provided to. Each drug is prescribed for 6 months. The symptom score check should be completed at the first outpatient visit(3 months after administration). We will Check the following items through abdominal ultrasound examination 6 months after administration.

: Gallbladder wall thickening presence and extent, number of gallstones, maximum diameter of gallstones, presence or absence of sludge. The general blood test (CBD) and general chemical test (SMA) are conducted three times at the first outpatient visit(3 months after administration), and the research expenses for 3 months and 6 months are supported by the research fund. In the final analysis, we compare the symptom scores between the two groups through the Student T-test, and compare the blood test and ultrasound using the Chi-square test. We want to confirm the following three things through this study. ① In patients with cholelithiasis with symptoms of dyspepsia, prospective data on the degree of symptom improvement following motilitone administration can be obtained. ② It is possible to evaluate the degree of relief or exacerbation of gallstones through ultrasound examination. ③ It is expected that it will be effective in improving symptoms and alleviating cholelithiasis in patients with dyspeptic cholelithiasis due to increased gallbladder contractility of motilitone.

ELIGIBILITY:
Inclusion Criteria:

1. 19 years old to under 75
2. Patients with dyspepsia in patients with cholelithiasis
3. Patients who consented to this study and conducted questionnaires and tests during follow up

Exclusion Criteria:

1. asymptomatic cholelithiasis
2. Gallstones over 3cm
3. Acute cholecystitis requires surgery
4. pregnant women
5. porcelain gallbladder
6. Chronic cholecystitis with severe thickening of the gallbladder wall
7. Patients with anomalous pancreato-biliary duct union,
8. When other physicians believe that surgery is necessary
9. Patients with a history of hypersensitivity to "motilitone" or its components

   ; Since this drug contains lactose, galactose intolerance, Patients with genetic problems such as Lapp lactase deficiency or glucose-galactose malabsorption.
10. Hepatitis patients (Hepatitis carriers, cirrhosis patients) or suspected liver failure (AST, ALT levels are 1.5 times or more of normal values)

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-03-25 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Check symptom improvement | 3months (At the first outpatient visit 3months after administration)
  The symptom score check should be completed at the first outpatient visit 3 months after administration. Nepean Dyspepsia Index- Korean version will be used to check the patient's indigestion symptoms. The questionnaire contains the following gastrointestinal symptoms How often it happened / how severe the symptoms were / how much it bothered you There are five (or six) answers. Gastrointestinal symptoms included Abdominal pain, Abdominal discomfort, Having a sour stomach, Heart burn, A Spasm of the stomach, Chest pain, Early fullness, Gastric acid reflux, Satiety after eating, pressure in the upper abdomen, Bloating of the upper abdomen, Nausea, Vomiting, Burp, Hard to breathe. The answer can be selected in 5 (6) numbers; from 0 to 4 (5). We will check the total score with the sum of each score. The symptom score is compared before and 3 months after administration.
Changes in serum concentrations of WBC count (10^3/µL), before and after the administration | 3months (At the first outpatient visit 3months after administration)
Changes in serum concentrations of RBC count (10^6/µL), before and after the administration | 3months (At the first outpatient visit 3months after administration)
Changes in serum concentrations of Hemoglobin (g/dL), before and after the administration | 3months (At the first outpatient visit 3months after administration)
Changes in serum concentrations of BUN (mg/dL), before and after the administration | 3months (At the first outpatient visit 3months after administration)
Changes in serum concentrations of Glucose (mg/dL), before and after the administration | 3months (At the first outpatient visit 3months after administration)
Changes in serum concentrations of Albumin (g/dL), before and after the administration | 3months (At the first outpatient visit 3months after administration)
Changes in serum concentrations of Total bilirubin (mg/dL), before and after the administration | 3months (At the first outpatient visit 3months after administration)
Changes in serum concentrations of Direct bilirubin (mg/dL), before and after the administration | 3months (At the first outpatient visit 3months after administration)
Changes in serum concentrations of Amylase (U/L), before and after the administration | 3months (At the first outpatient visit 3months after administration)
Changes in serum concentrations of Lipase (U/L), before and after the administration | 3months (At the first outpatient visit 3months after administration)
Changes in serum concentrations of Sodium (mmol/L), before and after the administration | 3months (At the first outpatient visit 3months after administration)
Changes in serum concentrations of Potassium (mmol/L), before and after the administration | 3months (At the first outpatient visit 3months after administration)
Changes in serum concentrations of liver enzymes (aspartate aminotransferase and alanine aminotransferase (IU/L)), before and after the administration | 3months (At the first outpatient visit 3months after administration)
Changes in serum concentrations of Alkaline phosphate (IU/L), before and after the administration | 3months (At the first outpatient visit 3months after administration)
Changes in serum concentrations of Gamma-glutamyltransferase (IU/L), before and after the administration | 3months (At the first outpatient visit 3months after administration)

SECONDARY OUTCOMES:
Abdominal ultrasound examination - Change of Gallbladder wall thickening | 6months (At the second outpatient visit 6months after administration)
  We will check Abdominal ultrasound examination 6months after administration. Ultrasonography checks whether the gallbladder wall is thick or not. The ultrasound findings are compared before and 6 months after administration.
Abdominal ultrasound examination - Gallbladder wall extent | 6months (At the second outpatient visit 6months after administration)
  We will check Abdominal ultrasound examination 6months after administration. If the gallbladder wall was thick at the first visit, ultrasound after 6 months checks how thick the gallbladder wall is. The thickness of the gallbladder wall is confirmed by mm from ultrasound findings. The ultrasound findings are compared before and 6 months after administration.
Abdominal ultrasound examination - Number of gallstones | 6months (At the second outpatient visit 6months after administration)
  We will check Abdominal ultrasound examination 6months after administration. Ultrasonography checks the number of gallstones. The ultrasound findings are compared before and 6 months after administration.
Abdominal ultrasound examination - Maximum diameter of gallstones | 6months (At the second outpatient visit 6months after administration)
  We will check Abdominal ultrasound examination 6months after administration. Ultrasonography checks the maximum diameter of gallstones. The maximum diameter of gallstones is confirmed by mm from ultrasound findings. The ultrasound findings are compared before and 6 months after administration.
Abdominal ultrasound examination - Presence or Absence of sludge | 6months (At the second outpatient visit 6months after administration)
  We will check Abdominal ultrasound examination 6months after administration. Ultrasonography checks whether the sludge is in the gallbladder or not. The ultrasound findings are compared before and 6 months after administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Severance hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Catnach SM, Ballinger AB, Stevens M, Fairclough PD, Trembath RC, Drury PL, Watkins PJ. Erythromycin induces supranormal gall bladder contraction in diabetic autonomic neuropathy. Gut. 1993 Aug;34(8):1123-7. doi: 10.1136/gut.34.8.1123. PMID 8174966
- [Background] Sengupta S, Modak P, McCauley N, O'Donnell LJ. Prokinetic effect of alpha-adrenergic antagonist, and beta-adrenergic antagonist on gall-bladder motility in humans with gall-stone disease. Eur J Gastroenterol Hepatol. 2007 Jul;19(7):581-3. doi: 10.1097/MEG.0b013e32811ec044. PMID 17556905